CLINICAL TRIAL: NCT00794170
Title: I-SIGHT: Interactive Study to Increase Glaucoma adHerence to Treatment Phase 2: Participant Recruitment & Intervention Delivery and Evaluation
Brief Title: Interactive Study to Increase Glaucoma Adherence to Treatment
Acronym: I-SIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Karen Glanz, MD, Adjunct Professor of Public Health, Emory University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB00001335; R01EY016997 (NIH); I-SIGHT (Other: Other)
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: Treatment Compliance
MeSH Terms: conditions — Glaucoma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone and print based intervention (Experimental): The I-SIGHT intervention consists of twelve interactive voice recognition (IVR) phone calls over a nine-month period and accompanying printed materials that are mailed to participants following each call. The phone call messages and print materials are tailored to individuals' circumstances using data from the screening and baseline interviews. The intervention is based on theoretical constructs from Social Cognitive Theory and the Health Belief Model, and emphasizes self-efficacy, medication taking skills, outcome expectancies, facilitators and barriers to compliance, and social support. The treatment group receives the tailored telephone intervention and mailed, printed materials.
  Interventions: Behavioral: Telephone and Print based intervention
- Usual care (No Intervention): The control group received usual care at each clinical site and interacted with study personnel only for data collection.

INTERVENTIONS:
Behavioral: Telephone and Print based intervention — Thiss intervention consisted of tailored phone calls and follow-up mailings.
  Arms: Telephone and print based intervention

SUMMARY:
Study participants who receive the I-SIGHT intervention will have higher rates of glaucoma treatment compliance (e.g., medication-taking and refill compliance, return for clinical follow-up) and more positive eye health outcomes at 12-month follow-up than participants who receive the control group intervention.

DETAILED DESCRIPTION:
The intervention is telephone-based and individually-tailored to participants' compliance knowledge, attitudes, and behaviors; psychosocial predictors of compliance; health literacy; race and culture; and prescribed medication regimen. The intervention calls utilize interactive voice recognition technology to facilitate interest, participation, and interaction with call recipients. We evaluated the intervention in a randomized controlled trial with telephone interviews administered to all participants at baseline, 6, 9, and 12-months

ELIGIBILITY:
Inclusion Criteria:

* Receive treatment at the Atlanta VA Medical Center or Grady Eye clinic for their eye condition
* Be between the ages of 18-80
* Be Caucasian or African American
* Possess a telephone (home telephone or cellular phone)
* Speak and understand English
* Be diagnosed with open angle glaucoma, be glaucoma suspect, or be ocular hypertensive for at least one year
* Be prescribed daily doses of topical treatments for at least one year
* Be able to read or have someone who can help the participant with reading written materials that we give to the participant

Exclusion Criteria:

* Having eye surgery within 3 months of baseline interview and enrollment
* Being legally blind (20/200 or worse)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia

REFERENCES:
- [Derived] Glanz K, Beck AD, Bundy L, Primo S, Lynn MJ, Cleveland J, Wold JA, Echt KV. Impact of a health communication intervention to improve glaucoma treatment adherence. Results of the interactive study to increase glaucoma adherence to treatment trial. Arch Ophthalmol. 2012 Oct;130(10):1252-8. doi: 10.1001/archophthalmol.2012.1607. PMID 22688429

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone and Print Based Intervention: The I-SIGHT intervention consists of twelve interactive voice recognition (IVR) phone calls over a nine-month period and accompanying printed materials that are mailed to participants following each call. The phone call messages and print materials are tailored to individuals' circumstances using data from the screening and baseline interviews. The objectives of the calls are to provide individually-tailored messages to encourage compliance with medication taking, appointment-keeping, and refills (based on self-report); to provide knowledge about glaucoma; and to counsel patients on how to address barriers to compliance. The intervention is based on theoretical constructs from Social Cognitive Theory and the Health Belief Model, and emphasizes self-efficacy, medication taking skills, outcome expectancies, facilitators and barriers to compliance, and social support. The treatment group receives the tailored telephone intervention and mailed, printed materials.
- Usual Care: The control group receives usual care at each clinical site and interacts with study personnel only for data collection.
Period: Overall Study
Arm/Group | Telephone and Print Based Intervention | Usual Care
Started | 157 | 155
Completed | 150 | 152
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Telephone and Print Based Intervention: This was a tailored phone call followed up by print materials.
- Usual Care: control
- Total: Total of all reporting groups
Arm/Group | Telephone and Print Based Intervention | Usual Care | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 95 | 186
  >=65 years | 66 | 60 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 98 | 97 | 195
Region of Enrollment [Number; unit: participants]
  United States | 157 | 155 | 312

OUTCOME MEASURES:

1. Primary Outcome: Data on Prescription Drug Renewals, Appointment Compliance and Medication Taking (e.g. Physician Notes)
Description: The adherence measure, developed and pilot tested by the I-SIGHT study team, assessed compliance adherence with medication taking, refills, and appointment-keeping by self-report and chart review. Subjects were considered nonadherent with medication-taking if they reported missing doses of any glaucoma medication within one month of the interview. Levels of medication-taking nonadherence were also examined by missed doses within 7 days, 2 weeks, or 1 mo of the interview. Nonadherence with refills was defined as running out of any glaucoma medication and missing a dose within a specified time frame (i.e. 1 year prior to the baseline interview; 6 months prior to 6-month interview; and 3 months prior to the 9 and 12 month interview). Appointment-keeping nonadherence was indicated by self-report of missing a glaucoma treatment appointment and not rescheduling during the specified time frame. Self-report of nonadherence in any of these three areas classified the subject as nonadherent.
Time Frame: Baseline and 12 months
Population: The two treatment groups were compared on change in the percent of adherent patients between baseline and follow-up using a longitudinal logistic regression model fit using a generalized linear model. A p-value less than 0.05 was considered statistically significant. No statistical comparison was done.
Measure: Number; unit: participants
Groups:
- Telephone and Print Intervention: The I-SIGHT intervention consists of twelve interactive voice recognition (IVR) phone calls over a nine-month period and accompanying printed materials that are mailed to participants following each call. The phone call messages and print materials are tailored to individuals' circumstances using data from the screening and baseline interviews. The objectives of the calls are to provide individually-tailored messages to encourage compliance with medication taking, appointment-keeping, and refills (based on self-report); to provide knowledge about glaucoma; and to counsel patients on how to address barriers to compliance. The intervention is based on theoretical constructs from Social Cognitive Theory and the Health Belief Model, and emphasizes self-efficacy, medication taking skills, outcome expectancies, facilitators and barriers to compliance, and social support. The treatment group receives the tailored telephone intervention and mailed, printed materials.
- Usual Care: The control group receives usual care at each clinical site and interacts with study personnel only for data collection. Both groups receive birthday cards from the study team.
Arm/Group | Telephone and Print Intervention | Usual Care
Number analyzed (Participants) | 157 | 155
participants | 150 | 152

ADVERSE EVENTS:
Arm/Group | Telephone and Print Based Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/155
Other Adverse Events (participants affected / at risk) | 0/157 | 0/155

LIMITATIONS AND CAVEATS:
There may have been a selection bias that contributed to a placebo effect in the control group. The "control" patients may have already been motivated to seek knowledge or involvement in management of glaucoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No